CLINICAL TRIAL: NCT04365543
Title: Unified Protocol to Help Emotions and Promote Auditory Relief (U-HEAR).
Brief Title: Treatment for Youth (Ages 8 to 16 Years Old) With Misophonia (U-HEAR)
Acronym: U-HEAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Lewin, Associate Professor and Interim Division Chief, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro#00042498
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Misophonia
Keywords: misophonia; sensory sensitivity; anxiety; sound
MeSH Terms: conditions — misophonia; Anxiety Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP-C/A for Misophonia (Experimental): The Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents (UP-C/A) are manualized treatments for treating emotional disorders in youth. We have modified the UP-C/A to meet the needs for youth with misophonia.
  Interventions: Behavioral: Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents (UP-C/A) for youth with misophonia
- Psychoeducation and Relaxation Therapy (Experimental): Psychoeducation and Relaxation Therapy (PRT) is a treatment that educates the child on misophonia and provides training in relaxation skills and tools for calming panic, anxiety and anger feelings.
  Interventions: Behavioral: Psychoeducation and Relaxation Therapy (PRT)

INTERVENTIONS:
Behavioral: Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents (UP-C/A) for youth with misophonia — Please see arm/group descriptions
  Arms: UP-C/A for Misophonia
Behavioral: Psychoeducation and Relaxation Therapy (PRT) — Please see arm/group descriptions
  Arms: Psychoeducation and Relaxation Therapy

SUMMARY:
If someone is really sensitive to certain noises and sounds, they might have misophonia. U-HEAR is a study created to find out what helps kids and teens with misophonia. There are two treatments being tested in this study. The treatment your child receives will be determined at random. There will be a Two-Thirds (2/3rds or 66%) chance your child will receive a treatment called the Unified Protocol for Children and Adolescents (UP-C/A) that has been modified to meet the needs for youth with misophonia. There is a One-Third (1/3rd or 33%) chance your child will receive a treatment called Psychoeducation and Relaxation. All participants will get ten free treatment sessions. Each session will last one hour and happen once a week. The aim of the study is to evaluate the feasibility and preliminary efficacy of the UP-C/A for youth with misophonia.

DETAILED DESCRIPTION:
Misophonia is a condition characterized by intense affective and/or physical responses to auditory triggers. Negative affective states, including significant distress and avoidance are characteristic of misophonia. These negative emotional responses to trigger sounds, which result in behavioral problems and impairment, may be the primary targets for effective psychosocial intervention for misophonia. Transdiagnostic treatment approaches address clinically-significant distress through the use of evidence-based, cognitive-behavioral techniques (e.g., mindful awareness, problem-solving, and opposite action strategies) that allow for flexible and personalized treatment of core dysfunctions that cut across emotional disorders and lead to on-going impairment. This type of evidence-based, transdiagnostic approach includes skills applicable for problems observed frequently in misophonia including adaptability, problem solving, emotional (arousal) dysregulation and poor distress tolerance. The hypothesized mechanism of change of these core-dysfunction focused treatments is increased tolerance of distress in response to strong or intense emotion states. A secondary target is the reduction of maladaptive emotional behaviors (e.g., avoidance, aggression, escape) that may reinforce distress over time. To that end, this proposal aims to evaluate the feasibility and preliminary efficacy of the Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents (UP-C/A) for youth with misophonia. We will compare UP-C/A in a 2:1 ratio against a comparison condition (PRT: psychoeducation plus relaxation training), a behavioral approach that represents usual treatment in the community and has been utilized in clinical trials (35% response rate).

ELIGIBILITY:
Inclusion Criteria:

* The child meets criteria for misophonia
* The child is currently living with their family/guardian(s)
* The child is between 8 and 16 years old
* Parent/legal guardian and child are able to read and speak English without a translator
* Parent/legal guardian is able to attend weekly sessions and all assessments
* If the child is on a psychotropic medication, they will need to be on a stable dose for 4 weeks prior to assessment (2 weeks for stimulant medication)

Exclusion Criteria:

* The child has received prior UP-C/A treatment
* The child is acutely suicidal
* The child has a current diagnosis of psychosis, bipolar disorder, intellectual disability, alcohol/substance dependence, or eating disorder

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in symptoms measured by Clinical Global Impression - Improvement (5 weeks) | 5 weeks
  Clinical Global Impression-Improvement (CGI-I) is a 7-point clinician rated scale of treatment response anchored by 1 (very much improved) and 7 (very much worse). For categorical secondary outcomes, response is defined as a CGI-I rating of 1 or 2 (much improved/very much improved), and remission as CGI-S of 1 to 2. CGI-I will be used to measure symptom improvement after 5 weeks of treatment.
Improvement in symptoms measured by Clinical Global Impression - Improvement (10 weeks) | 10 weeks
  Clinical Global Impression-Improvement (CGI-I) is a 7-point clinician rated scale of treatment response anchored by 1 (very much improved) and 7 (very much worse). For categorical secondary outcomes, response is defined as a CGI-I rating of 1 or 2 (much improved/very much improved), and remission as CGI-S of 1 to 2. CGI-I will be used to measure symptom improvement after 10 weeks of treatment.
Severity of symptoms measured by Clinical Global Impression - Severity (Baseline) | Baseline
  Clinical Global Impression-Severity (CGI-S) is a widely used 7-point clinician rating of severity of psychopathology; raters will be instructed to score based on psychopathology and misophonia symptoms. Severity ratings range from 1 (no illness) to 7 (extremely severe). Severity will be measured before treatment begins to create a baseline for each participant.
Severity of symptoms measured by Clinical Global Impression - Severity (5 weeks) | 5 weeks
  Clinical Global Impression-Severity (CGI-S) is a widely used 7-point clinician rating of severity of psychopathology; raters will be instructed to score based on psychopathology and misophonia symptoms. Severity ratings range from 1 (no illness) to 7 (extremely severe). CGI-S will be used to measure severity after 5 weeks of treatment.
Severity of symptoms measured by Clinical Global Impression - Severity (10 weeks) | 5 weeks
  Clinical Global Impression-Severity (CGI-S) is a widely used 7-point clinician rating of severity of psychopathology; raters will be instructed to score based on psychopathology and misophonia symptoms. Severity ratings range from 1 (no illness) to 7 (extremely severe). CGI-S will be used to measure severity after 10 weeks of treatment.
Overall impairment measured by Child's Global Assessment Scale (Baseline) | Baseline
  Clinician rated measure of general functioning including impairment to capture functioning/impairment independent of diagnoses. The child or young person is given a single score between 1 and 100, based on a clinician's assessment of a range of aspects related to a child's psychological and social functioning. The score will put them in one of ten categories that range from 'extremely impaired' (1-10) to 'doing very well' (91-100. General functioning of the participant will be measured before treatment begins to create a baseline for each subject.
Overall impairment measured by Child's Global Assessment Scale (5 weeks) | 5 weeks
  Clinician rated measure of general functioning including impairment to capture functioning/impairment independent of diagnoses. The child or young person is given a single score between 1 and 100, based on a clinician's assessment of a range of aspects related to a child's psychological and social functioning. The score will put them in one of ten categories that range from 'extremely impaired' (1-10) to 'doing very well' (91-100). CGAS will be used to measure general functioning after 5 weeks of treatment.
Overall impairment measured by Child's Global Assessment Scale (10 weeks) | 10 weeks
  Clinician rated measure of general functioning including impairment to capture functioning/impairment independent of diagnoses. The child or young person is given a single score between 1 and 100, based on a clinician's assessment of a range of aspects related to a child's psychological and social functioning. The score will put them in one of ten categories that range from 'extremely impaired' (1-10) to 'doing very well' (91-100). CGAS will be used to measure general functioning after 10 weeks of treatment.

SECONDARY OUTCOMES:
Misophonia symptoms as measured by Misophonia Assessment Questionnaire | Baseline
  Misophonia Assessment Questionnaire (MAQ) is a 21 item, youth self-report, and parent-report questionnaire assessing severity and side effects of the youth's misophonia symptoms and reactions to misophonic sounds.
Change in misophonia symptoms as measured by Misophonia Assessment Questionnaire | 5 weeks
  Misophonia Assessment Questionnaire (MAQ) is a 21 item, youth self-report, and parent-report questionnaire assessing severity and side effects of the youth's misophonia symptoms and reactions to misophonic sounds.
Change in misophonia symptoms as measured by Misophonia Assessment Questionnaire | 10 weeks
  Misophonia Assessment Questionnaire (MAQ) is a 21 item, youth self-report, and parent-report questionnaire assessing severity and side effects of the youth's misophonia symptoms and reactions to misophonic sounds.
Misophonia symptoms as measured by Misophonia Questionnaire | Baseline
  The Misophonia Questionnaire is a 17-item questionnaire that assesses the presence of misophonia symptoms, emotions and behaviors associated with misophonic reactions, and symptom severity. The first two subscales are rated on a scale of 0 (not at all true) to 4 (always true). These two parts are summed to produce a total score ranging from 0 - 68. The severity subscale is a single item that asks an individual to provide a rating of their sound sensitivity on a scale from 0 (no sound sensitivities) to 15 (very severe sound sensitivities). The youth self-report (for those 10 and older) and parent report will serve as both a measure of symptoms of misophonia and allow for calculation of severity score.
Change in misophonia symptoms as measured by Misophonia Questionnaire | 5 weeks
  The Misophonia Questionnaire is a 17-item questionnaire that assesses the presence of misophonia symptoms, emotions and behaviors associated with misophonic reactions, and symptom severity. The first two subscales are rated on a scale of 0 (not at all true) to 4 (always true). These two parts are summed to produce a total score ranging from 0 - 68. The severity subscale is a single item that asks an individual to provide a rating of their sound sensitivity on a scale from 0 (no sound sensitivities) to 15 (very severe sound sensitivities). The youth self-report (for those 10 and older) and parent report will serve as both a measure of symptoms of misophonia and allow for calculation of severity score.
Change in misophonia symptoms as measured by Misophonia Questionnaire | 10 weeks
  The Misophonia Questionnaire is a 17-item questionnaire that assesses the presence of misophonia symptoms, emotions and behaviors associated with misophonic reactions, and symptom severity. The first two subscales are rated on a scale of 0 (not at all true) to 4 (always true). These two parts are summed to produce a total score ranging from 0 - 68. The severity subscale is a single item that asks an individual to provide a rating of their sound sensitivity on a scale from 0 (no sound sensitivities) to 15 (very severe sound sensitivities). The youth self-report (for those 10 and older) and parent report will serve as both a measure of symptoms of misophonia and allow for calculation of severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lewin, PhD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Child and Adolescent Mood and Anxiety Treatment (CAMAT) Program at the University of Miami, Coral Gables, Florida
  - University of Florida Rothman Center, St. Petersburg, Florida

IPD SHARING:
Plan to Share IPD: Yes
The sponsor requests de-identified data as a grant requirement in order to better the understand of misophonia. At the conclusion of the study, we will provide the de-identified data.
Supporting Information: Study Protocol, SAP
Time Frame: Approximately 2 years following the completion of the analyses. Duration of the availability is at Sponsor's discretion.
Access Criteria: Access is at Sponsor's discretion.